CLINICAL TRIAL: NCT03575897
Title: Serial Assessment of Body Fat Accrual in Very Preterm Infants: A Pilot Randomized Trial
Brief Title: Serial Assessment of Body Fat Accrual in Very Preterm Infants
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Ariel A. Salas, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 300001753; 2U54MD000502 (NIH)
Record Dates: First submitted 2018-06-21; First posted 2018-07-03 (Actual); Results first posted 2021-05-17 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Infant,Premature; Body Weight; Adiposity
Keywords: Premature Infants; Body composition
MeSH Terms: conditions — Premature Birth; Body Weight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Intervention Group (Experimental): Infants randomly assigned to the intervention group will undergo serial measurements of infant body composition during their hospitalization. This information about infant body composition will be known to the clinicians caring for them (including reference data).
  Interventions: Diagnostic Test: Assessment of infant body composition
- Control Group (Active Comparator): Infants randomly assigned to the control group will also undergo serial measurements of infant body composition during their hospitalization, but this information will not be available to the clinicians caring for them.
  Interventions: Diagnostic Test: Assessment of infant body composition

INTERVENTIONS:
Diagnostic Test: Assessment of infant body composition — Serial assessments of infant body composition with air displacement plethysmography in very preterm infants will occur in the first 14 days after birth (baseline measure), at 32 weeks postmenstrual age (PMA), and at 36 weeks PMA or hospital discharge (whichever occurs first)

SUMMARY:
Despite evidence that both rapid weight gain and excessive body fat accrual are associated with overweight and obesity, usual neonatal care of preterm infants does not include assessment of body fat accrual. The study hypothesis is that identification of early changes in infant body composition (i.e. amount of fat mass and fat-free mass) reduces % body fat at 3 months of age.

DETAILED DESCRIPTION:
Infants in the intervention group will have the information about infant body composition known to the clinicians caring for them (including reference data). Infants in the control group will also undergo serial measurements of infant body composition, but this information will not be available to the clinicians.

If parent agrees, stool "dirty" diapers will be collected 2 times (at the time of hospital discharge and at 3 months of corrected age).

ELIGIBILITY:
Inclusion Criteria:

* Gestational age between 28 and 32 weeks of gestation

Exclusion Criteria:

* Gastrointestinal or neurologic malformations
* Terminal illness requiring limited or withheld support

Ages: 1 Day to 14 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2020-01-16 (Actual); Study Completion 2025-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ariel A. Salas, MD, MSPH, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Result] Salas AA, Jerome ML, Chandler-Laney P, Ambalavanan N, Carlo WA. Serial assessment of fat and fat-free mass accretion in very preterm infants: a randomized trial. Pediatr Res. 2020 Nov;88(5):733-738. doi: 10.1038/s41390-020-1052-x. Epub 2020 Jul 7. PMID 32634820

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention Group | Control Group
Started | 25 | 25
Completed | 13 | 12
Not Completed | 12 | 13
Not completed — Lost to Follow-up | 12 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Control Group | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 25 | 25 | 50
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: Weeks] | 31 [30 to 32] | 30 [30 to 32] | 30 [30 to 32]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 14 | 24
  Male | 15 | 11 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 12 | 23
  White | 14 | 13 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Infant Body Composition
Description: Percent body fat estimated by air displacement plethysmography
Time Frame: Assessed at 3 months of corrected age
Measure: Mean (Standard Deviation); unit: percentage of body fat
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 12 | 13
percentage of body fat | 21 (4) | 19 (6)

2. Secondary Outcome: Growth
Description: Weekly weight gain in grams
Time Frame: Birth to 3 months of corrected age
Measure: Median (Inter-Quartile Range); unit: grams/kg/day
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 13 | 12
grams/kg/day | 8 [7 to 9] | 9 [7 to 9]

3. Secondary Outcome: Length
Description: Length in cm at 3 months of corrected age
Time Frame: 3 months of corrected age
Population: 2 infants in the control group did not have a length measurement at 3 months of corrected age
Measure: Median (Inter-Quartile Range); unit: cm
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 13 | 10
cm | 59 [56 to 60] | 60 [57 to 62]

4. Secondary Outcome: Head Circumference
Description: Head circumference in cm at 3 months of corrected age
Time Frame: 3 months of corrected age
Measure: Median (Inter-Quartile Range); unit: cm
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 12 | 10
cm | 40 [39 to 42] | 41 [40 to 42]

5. Secondary Outcome: Body Mass Index
Description: Weight and height at 3 months of corrected age combined to report BMI in kg/m^2
Time Frame: 3 months of corrected age
Measure: Median (Inter-Quartile Range); unit: kg/m^2
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 13 | 12
kg/m^2 | 5 [4 to 6] | 6 [5 to 6]

6. Secondary Outcome: Infant Body Composition
Description: Percent body fat estimated by air displacement plethysmography
Time Frame: Assessed at 36 weeks of postmenstrual age or hospital discharge (whichever occurs first)
Measure: Mean (Standard Deviation); unit: percentage of body fat
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 18 | 17
percentage of body fat | 14 (5) | 14 (3)

7. Other Pre Specified Outcome: Changes in Intestinal Microbiome
Description: Determined by molecular analyses of bacteria in fecal samples
Time Frame: Birth to 3 months of corrected age
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Changes in Metabolic Pathways
Description: Determined by molecular analyses of serum samples
Time Frame: Birth to 3 months of corrected age
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Intervention Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-14): https://cdn.clinicaltrials.gov/large-docs/97/NCT03575897/Prot_SAP_001.pdf